## Evaluation of Gingival Crevicular Fluid and Saliva SOST and TWEAK, Gingival Crevicular Fluid RANKL and OPG Levels in Smokers and Non-smokers with Periodontitis

14.09.2023

## INFORMED CONSENT FORM - BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU Tarih / Versiyon Sayfa TİTCK-KAD-D2 05.05.2019 / Ver3.0 1/3

Çalışmanın Adı: Dişeti Oluğu Sıvısı ve Tükürük SOST ve TWEAK Dişeti Oluğu Sıvısı RANKL ve OPG Seviyelerinin Sigara İçen ve İçmeyen Periodontitisli Hastalarda Değerlendirilmesi

Sayın gönüllü,

Gazi Üniversitesi Diş Hekimliği Fakültesi Periodontoloji Anabilim Dalında Dt. Ece Güner tarafından yürütülen yukarıda adı verilen tez çalışmasına katılmak üzere davet edilmiş bulunuyorsunuz. Bu araştırmaya katılım tamamen gönüllük esasına dayanmaktadır. Bu çalışmanın sonuçları bilimsel amaçlarla kullanılacaktır. Çalışmadan çekilmeniz ya da araştırmacı tarafından çalışmadan çıkarılmanız halinde, sizle ilgili veriler kullanılmayacaktır. Ancak veriler bir kez anonimleştikten sonra çalışmadan çekilmeniz mümkün olmayacaktır. Sizden elde edilen tüm bilgiler gizli tutulacak, çalışma yayınlandığında da varsa kimlik bilgilerinizin gizliliği korunacaktır. Çalışmaya katılmanız durumunda herhangi bir mali yük altına girmeyeceksiniz ve size de herhangi bir ödeme yapılmayacaktır. Bu çalışmada yer almayı kabul etmeden önce, çalışmanın ne amaçla yapılmak istendiğini anlamanız ve kararınızı bu bilgilendirme çerçevesinde özgürce vermeniz gerekmektedir. Aşağıdaki bilgileri lütfen dikkatlice okuyunuz, sorularınız olursa sorunuz ve açık yanıtlar isteyiniz.

Çalışmanın amacı; sigara kullanımının dişeti hastalığı üzerine etkisini sigara kullanan ve sigara kullanmayan dişeti hastalığına sahip bireylerde karşılaştırmaktır. Çalışmaya Gazi Üniversitesi Diş Hekimliği Fakültesi Periodontoloji Anabilim Dalına kontrol ya da tedavi amaçlı başvuran, 18-70 yaş aralığındaki 78 gönüllü dahil edilecektir. Çalışmaya katılmayı kabul eden gönüllüler; periodontitis teşhisi konan sigara içmeyen, periodontitis teşhisi konan, sigara içen ve periodontal olarak sağlıklı, sigara içmeyen olarak üç gruba ayrılacaktır. Çalışmaya katılmayı kabul eden gönüllülerden dişeti hastalığının düzeyini belirlemek için rutin klinik ölçümler yapılacak, dişeti ve diş arasında bulunan aralıktaki sıvı ve tükürük toplanacaktır. Katılımcılardan alınacak kinik ölçümler için klinikte kullanılan rutin bir sond kullanılacaktır. Dişeti ve diş arasında bulunan aralıktaki sıvıyı toplamak için sıvıyı emen, ince, kağıt şeritler kullanılacak ve sıvıyı toplamak için kağıt şeritler dişeti ve diş arasındaki aralığa yerleştirilecektir. Katılımcılar tükürük toplanması için, bir bardağa 5 dakikalık süreç içerisinde ağızlarında biriken tükürüğü tüküreceklerdir. Yapılacak ölçümlerden ve sıvı örneği alma işlemlerinden sonra şişlik, ağrı, kanama, enfeksiyon gibi komplikasyonlar beklenmemektedir. Gönüllüler çalışmaya katılmayı kabul ettikten sonra ölçümler yapılacak ve sıvı örneklerinin toplanması tamamlandıktan sonra çalışma sonlanacaktır. Toplanan sıvı örnekleri Gazi Üniversitesi Tıp Fakültesi İmmünoloji Anabilim Dalında incelenecektir.

"Yukarıda yer alan ve çalışmaya başlanmadan önce gönüllülere verilmesi gereken bilgileri içeren metni okudum (ya da sözlü olarak dinledim). Eksik kaldığını düşündüğüm konularda sorularımı araştırmacılara sordum ve doyurucu yanıtlar aldım. Yazılı ve sözlü olarak tarafıma sunulan tüm açıklamaları ayrıntılarıyla anladığım kanısındayım. Çalışmaya katılmayı isteyip istemediğim konusunda karar vermem için yeterince zaman tanındı.

| Bu koşullar altında, çalışma kapsamında elde edilen şahsıma ait bilgilerin bilimsel amaçlarla kullanılmasırı gizlilik kurallarına uyulmak kaydıyla sunulmasını ve yayınlanmasını, hiçbir baskı ve zorlama altınd kalmaksızın, kendi özgür irademle kabul ettiğimi beyan ederim." |
|---|
| Gönüllünün Adı Soyadı: |
| İmza: |
| Tarih: 14.09.2023 |
| Araştırmacının Adı Soyadı: |
| İmza: |
| Tarih: |